CLINICAL TRIAL: NCT00503555
Title: Creation of a PBRN to Study Healthcare Delivery to a Transitioning Community
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Agency for Healthcare Research and Quality (AHRQ) (U.S. Federal Agency)
Other Study IDs: 1R03HS016023-01 (AHRQ)
Record Dates: First submitted 2007-07-17; First posted 2007-07-18 (Estimated); Last update posted 2007-08-30 (Estimated); Status verified 2006-10

CONDITIONS: Health Care Quality, Access, and Evaluation
Keywords: Primary Health Care; Hispanic Americans

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Other

SUMMARY:
The purpose of this study is the creation of a PBRN that will comprise primary care providers, community health organizations, community advocates and a research core of two academic institutions in order to study the healthcare needs of a rapidly growing immigrant population.

DETAILED DESCRIPTION:
The Carolinas Healthcare System (CHS) Department of Family Medicine in partnership with The University of North Carolina at Charlotte (UNCC) Geography Department have initiated a primary-care practice-based research network (PBRN) bringing together primary care physicians, local academic centers, and community organizations to study healthcare delivery to the burgeoning Hispanic population in Charlotte, North Carolina. CHS has created six primary care ambulatory clinics that serve as teaching centers and as "safety-net" practices for disadvantaged patients within the community. Despite many similarities between the clinics, including a shared informatics system, no research network currently exists. Creation of the proposed PBRN would allow the participating primary care providers to evaluate the community they serve, determine disparities in healthcare access and delivery, and to elucidate the impact of current services on the community. In addition, the PBRN brings together two academic institutions with prior experience implementing the community-oriented primary care model and the use of Geographic Information Systems tools for evaluating communities and understanding health care access.

The neighborhoods surrounding the CHS clinics have changed drastically over the past two decades secondary to a marked increase in Hispanic immigration to the area. This growth has produced an increasing demand on local healthcare providers. Our goal is to utilize the newly created research network to better understand healthcare delivery to the transitioning Hispanic population and thereby maximize quality of care and the efficacy of its delivery. Community organizations will be involved from the outset to allow community-based participation in the research design and overall goals. Creation of this initial PBRN will be used to lay the groundwork for expansion into other primary care practices and to seek funding for further research initiatives to improve community health.

ELIGIBILITY:
Inclusion Criteria:

* Hispanic

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 2006-06; Study Completion 2006-10 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Dulin, MD, PhD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Carolinas Medical Center - Eastland, Charlotte, North Carolina, United States

REFERENCES:
- See also: Official study webpage — http://www.carolinasmedicalcenter.org/body.cfm?id=1219&oTopID=0